CLINICAL TRIAL: NCT03149978
Title: Tumor Response Prediction in Neoadjuvant Chemoradiation of Locally Advanced Rectal Cancer Using Metabonomics Analysis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zhu Ji (Other)
Responsible Party: Sponsor-Investigator, Zhu Ji, Professor, Fudan University
Organization: Fudan University (Other)
Other Study IDs: FDRT-006
Record Dates: First submitted 2017-05-09; First posted 2017-05-11 (Actual); Last update posted 2017-05-12 (Actual); Status verified 2017-05

CONDITIONS: Locally Advanced Rectal Cancer
Keywords: Neoadjuvant Chemoradiation; treatment effect prediction; metabonomics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, plasma，serum and urine
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study suggested an effective application of pattern recognition, which figured the possible biological function of potential bio-markers of rectal cancer found in our study based on their chemical structures. Hence, this study identified the precursor protein and metabolic mechanism of these bio-markers and may contribute to the neoadjuvant chemoradiation of locally advanced rectal cancer

ELIGIBILITY:
Inclusion Criteria:

1. history of primary rectal cancer with distance from anal verge being less than 12 cm;
2. histologically confirmed adenocarcinoma;
3. initial pathological stage of T3 or T4 and/or N+;
4. no history of initial distant metastases;
5. Karnofsky Performance Status score of ≥75
6. ≥18 years;≤75 years
7. sign the inform consent

Exclusion Criteria:

1. pregnancy or breast-feeding women
2. serious medical illness
3. baseline blood and biochemical indicators do not meet the following criteria: neutrophils≥1.5×10^9/L, Hb≥90g/L, PLT≥100×10^9/L, ALT/AST ≤2.5 ULN, Cr≤ 1 ULN

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stage T3 or T4 and/or N+ rectal adenocarcinoma cancer eligible for neoadjuvant chemoradiation
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2014-07-01; Primary Completion 2017-12-30 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
TRG | Surgery scheduled 6-8 weeks after the end of chemoradiation
  Tumor regression grade

SECONDARY OUTCOMES:
Pathologic Complete Response | Surgery scheduled 6-8 weeks after the end of chemoradiation
Local Control rate | From date of randomization until the date of first documented pelvic failure, assessed up to 10 years
  Number of participants with pelvic failure after surgery, evaluated using Kaplan-Meier Curve
Disease-free Survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 10 years
Overall Survival | From date of randomization until the date of death from any cause, assessed up to 10 years
Number of participants with chemoradiation-related adverse events as assessed by CTCAE v4.0 | Up to 2 years
  Number of participants with chemoradiation-related adverse events as assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital, Fudan University, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Jia H, Shen X, Guan Y, Xu M, Tu J, Mo M, Xie L, Yuan J, Zhang Z, Cai S, Zhu J, Zhu Z. Predicting the pathological response to neoadjuvant chemoradiation using untargeted metabolomics in locally advanced rectal cancer. Radiother Oncol. 2018 Sep;128(3):548-556. doi: 10.1016/j.radonc.2018.06.022. Epub 2018 Jul 2. PMID 30041962